CLINICAL TRIAL: NCT05434871
Title: The Efficacy of Yoga in Pediatric Cancer Patients: A Randomized Controlled Study
Brief Title: Yoga in Pediatric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK-320
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Pediatric Cancer
Keywords: Pediatric Cancer; Yoga; Physiotherapy; Quality of Life; Fatigue; Pain; Motor Proficiency
MeSH Terms: conditions — Neoplasms; Fatigue; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): There will be a 45-minute yoga session 2 days a week for 8 weeks. Warm up with yoga-specific moves for 10 minutes (light stretching), yoga postures for 25 minutes and rest and meditate for the last ten minutes.
  Interventions: Other: Yoga training
- Control Group (Active Comparator): The routine physiotherapy and rehabilitation program consists of strength, flexibility, balance, gait and coordination exercises 2 days a week for 8 weeks.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Yoga training — There will be a 45-minute yoga session 2 days a week for 8 weeks. Warm up with yoga-specific moves for 10 minutes (light stretching), yoga postures for 25 minutes and rest and meditate for the last ten minutes.
  Arms: Yoga Group
Other: Physiotherapy — The standard physiotherapy and rehabilitation program consists of strength, flexibility, balance, gait and coordination exercises 2 days a week for 8 weeks.
  Arms: Control Group

SUMMARY:
Pediatric cancer patients and their families experience biopsychosocial difficulties as a result of the long and difficult treatment procedure, which have a severe impact on their quality of life. These difficulties might arise as a result of cancer and its treatment. Fatigue, pain, and an impaired motor skills are all common issues. These issues result in body structure and function deficits, as defined by the International Classification of Functioning-Child and Youth (ICF-CY), and have a negative impact on children's activity and participation levels. Yoga is a form of exercise that incorporates breathing methods, physical postures, and meditation. Yoga appears to relieve fatigue and improve quality of life in pediatric cancer patients, according to preliminary studies. However, no randomized controlled trial has been conducted in this population to determine the effectiveness of yoga. The purpose of this study is to assess children's quality of life, fatigue, pain, motor proficiency, participation, coping, and motivation; also to look at the effects of parents on quality of life, depression, fatigue, and care burden in a randomized controlled study.

DETAILED DESCRIPTION:
Childhood cancers are diseases that affect children and their families worldwide and occur in a variety of diagnostic groups. The focus has been on reducing mortality rates and long-term survival expectations in pediatric cancer patients, as well as reducing long-term side effects and improving quality of life, and it has become critical to develop interventions for problems that have long-term consequences. Within the framework of ICF-CY, biological problems such as exhaustion, pain, nausea, vomiting, and sleep difficulties, which are the most common symptoms in pediatric cancer patients, are included in body structure and function disorders. However, rather than cancer, the underlying cause of many difficulties is considered to be the treatment process itself. The symptoms experienced by pediatric cancer patients are moderate to high and are related to the stress level of the parents. As a result, improvements in pediatric cancer patients' symptoms may also lower the burden of care for their parents. Within the scope of the ICF-CY model, these biopsychosocial difficulties encountered by the child and family are interrelated and have an impact on the child's and family's quality of life. Limitations of normal joint movement, contractures, muscle weakness, diminished flexibility and functional mobility, balance and gait problems are among the physical and functional performance deficits reported by pediatric cancer patients as a result of the disease and therapy. Physical disabilities have a negative impact on children's participation in daily activities and their quality of life. As a result, specific therapy strategies aimed at improving children's physical limitations are required. In the current systematic review, it was stated that exercise applied to pediatric cancer patients had positive effects on fatigue, muscle strength, functional mobility, flexibility, sleep, physical activity level, and quality of life. No side effects were observed in the studies. In a meta-analysis, it was found that exercise, regardless of the type of exercise, lowers fatigue in pediatric cancer patients. Yoga is one of the promising approaches for children with cancer. Yoga improves stress and anxiety management, motor performance, concentration ability, and cardiovascular and musculoskeletal system functions in healthy children. Researchers reviewed yoga therapy in adult and pediatric cancer patients. Although yoga has been shown to improve psychological and physical functions in adults with cancer, the same cannot be said for children with cancer. In the literature, there are very few research on the impact of yoga on children with cancer. Children and their parents noted that after practicing yoga, sickness, the need for painkillers, and anxiety levels decreased, while sleep and mood improved. Yoga was useful in reducing stress and anxiety, according to the children and parents. In the existing literature, however, studies exploring the benefit of yoga in pediatric cancer patients are both quantitatively and qualitatively limited. In the literature, there is no randomized controlled trial that looks at the efficacy of yoga in children with cancer. The number of investigations in the literature is restricted to only eight pilot studies. This study is aimed to investigate the effects of yoga on quality of life, fatigue, pain, motor proficiency, and motivation in pediatric cancer patients in order to fill this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a hematological malignancy or a solid tumor
* Age between 6 years and 12 years
* Received chemotherapy for at least two weeks
* Ability to stand and move without the use of an assistive device
* To be able to read and speak Turkish

Exclusion Criteria:

* Diagnosis of central nervous system tumor, genetic syndrome or neurological disorder
* Surgery planned within the 8-week period planned to participate in yoga
* Refused to participate the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQL) Cancer Module | change from baseline to end of the 8 weeks
  The PedsQL-Cancer Module assesses the quality of life and symptoms of children diagnosed with pediatric cancer. Both the parent and child versions of the PedsQL-Cancer Module are available. The scale contains 26 items divided into eight domains: pain (2 items), nausea (5 items), operational anxiety (3 items), treatment anxiety (3 items), anxiety (3 items), cognitive issues (4 items), perceived physical appearance (3 items), and communication (3 items). It can be used on children with pediatric cancer aged 2-4, 5-7, and 8-12 years old. Minimum score is 0 and maximum score is 100.
Child Fatigue Scale-R 24-Hours | change from baseline to end of the 8 weeks
  The Child Fatigue Scale-24 Hour (CFS-24 hours) is a scale that measures how tired children aged 7 to 12 were in the previous 24 hours. There are child and parent versions of CFS-24 hours. The CFS-24 child form contains 10 items. Each item is scored on a 5-point Likert scale. It is rated as 1 = not at all and 5 = very much. The scale total score is classified between 10 = no fatigue and 50 = high fatigue.
Pain Flexibility Scale for Children with Cancer | change from baseline to end of the 8 weeks
  The scale assesses children's pain acceptance in chronic pain.It has a total of 20 questions divided into two sub-sections: valued activities and pain resistance. Pain resistance examines pain avoidance and control, whereas valued behaviors assesses involvement in meaningful activities despite pain. The scale is a seven-point Likert scale, with 0 indicating total disagreement (never true), and 6 indicating total agreement (Always true).
Bruininks-Oseretsky Test of Motor Proficiency Short Form -BOT-2 SF: | change from baseline to end of the 8 weeks
  The Bruininks-Oseretsky Test of Motor Proficiency is a norm-referenced test. The Bruininks-Oseretsky Test of Motor Proficiency is a test that evaluates children's gross and fine motor skills between the ages of 4 and 21. It evaluates four different aspects of motor skills: fine manual control, manual coordination, body coordination, strength, and agility. Long and short versions are available. The short form comprises 14 items and contains some of the items from the long form. The results of the The Bruininks-Oseretsky Test of Motor Proficiency Short Form are given as standard scores or percentiles. In addition, outcomes may be classified as below average or above average in a descriptive category. Minimum point score is 0 and maximum point score is 88.
Pediatric Motivation Scale | change from baseline to end of the 8 weeks
  PMOT assesses the motivation of children ages 8 to 18 to participate in a rehabilitation program. There are 21 items in total, divided into six categories: effort-importance, interest-enjoyment, competence, relatedness, autonomy, and value-usefulness. The first 19 questions are answered using a six-point smiley face scale (1 = not true at all, 6 = definitely true). The questions 20 and 21 are also open-ended. More motivation is indicated by higher scores.
Paediatric Cancer Coping Scale | change from baseline to end of the 8 weeks
  For children aged 7-18 years, PCCS assesses children's notifications of cancer coping techniques. Cognitive coping, problem-focused coping, and defensive coping are the three subscales that comprise the PCCS. There are 33 items total. A likert scale with 0-3 points is used for scoring. From 0 to 99, the total rating is calculated. The higher the score, the better the coping ability.
Participation and Environment- Children and Youth (PEM-CY) | change from baseline to end of the 8 weeks
  PEM-CY is a parent-report questionnaire to assess participation and environment factors in the home, at school and within community settings. The participation sections included 10 activities in the home setting, five activities in the school setting and 10 in the community setting. For each activity, parents are asked to determine the participation frequency (how frequently has the child participated with eight options: daily to never), participation involvement (how involved the child is while participating the activity rated on a five-point scale: very involved to minimally involved) and whether change is desired (do the parents want to see change in the child's participation in this type of activity: no or yes, with 5 different types of change)
The Child Fatigue Scale-Parent Form | change from baseline to end of the 8 weeks
  The Child Fatigue Scale-Parent Form contains 17 items. It is scored on a 5-point Likert scale. The total score is classified between 17 = no fatigue and 85 = high fatigue.

SECONDARY OUTCOMES:
Nottingham Health Profile | change from baseline to end of the 8 weeks
  Nottingham Health Profile assess the physical, emotional and health problems perceived by a person. It consist of 6 different subcategories such as energy, pain, physical mobility, sleep, emotional reactions and social isolation with 38 items. Nottingham Health Profile examines that current state of health condition and the answers are dichotomous (yes/no). The overall value is calculated by multiplying the intensity of the questions by the positive answer to each one. The minimum score is 0, maximum score is 100.
Beck Depression Inventory (BDI) | change from baseline to end of the 8 weeks
  The BDI assesses characteristic attitudes and depression symptoms with 21 self-reported items. It takes about 10 minutes to finish the assessment. It is intended for people aged 13 and up. BDI includes 21 questions. For each question, the lowest score is 0 and the maximum score is 3. The total score of all answers is evaluated as follows 0 to 9 points: "minimal depressive symptoms", 10 to 16 points: "mild depressive symptoms", 17 to 29 points: "moderate depressive symptoms", 20 to 63 points: "severe depressive symptoms".
Fatigue Impact Scale | change from baseline to end of the 8 weeks
  It is a multidimensional scale that measures the physical, cognitive and social effects of fatigue. It consists of 40 items divided into 10 cognitive, 10 physical, and 20 social subscales. Each question is scored on a five-point Likert scale from 0 (no problem) to 4 (extreme problem). The maximum total point is 160.
The Fatigue Severity Scale | change from baseline to end of the 8 weeks
  The fatigue severity scale is the one of the most used scale that assess fatigue. There are nine questions. Each question is scored on a seven-point Likert scale from one to seven. The mean of nine questions is the scale value. Higher scores indicating more severe fatigue. Although there is no recommendation, it is usually considered that fatigue above 4 points is significant.
Caregiving Burden Scale for Family Caregivers of Children with Cancer-CBSFC-CC | change from baseline to end of the 8 weeks
  It assesses the burden of care of family members caregivers aged 0 to 18 who have been diagnosed with cancer. The measure assesses the burden of care in terms of physical, emotional, mental, socio-cultural, and economic factors over 36 items. The CBSFC-CC is measured on a 5-point Likert scale, with 1 indicating never and 5 indicating always.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results will be submitted to the journal.

REFERENCES:
- [Result] Tanner L, Keppner K, Lesmeister D, Lyons K, Rock K, Sparrow J. Cancer Rehabilitation in the Pediatric and Adolescent/Young Adult Population. Semin Oncol Nurs. 2020 Feb;36(1):150984. doi: 10.1016/j.soncn.2019.150984. Epub 2020 Jan 24. PMID 31983485
- [Result] Hooke MC, Linder LA. Symptoms in Children Receiving Treatment for Cancer-Part I: Fatigue, Sleep Disturbance, and Nausea/Vomiting. J Pediatr Oncol Nurs. 2019 Jul/Aug;36(4):244-261. doi: 10.1177/1043454219849576. PMID 31307321
- [Result] Linder LA, Hooke MC. Symptoms in Children Receiving Treatment for Cancer-Part II: Pain, Sadness, and Symptom Clusters. J Pediatr Oncol Nurs. 2019 Jul/Aug;36(4):262-279. doi: 10.1177/1043454219849578. PMID 31307323
- [Result] Olagunju AT, Sarimiye FO, Olagunju TO, Habeebu MY, Aina OF. Child's symptom burden and depressive symptoms among caregivers of children with cancers: an argument for early integration of pediatric palliative care. Ann Palliat Med. 2016 Jul;5(3):157-65. doi: 10.21037/apm.2016.04.03. Epub 2016 May 9. PMID 27199271
- [Result] Svavarsdottir EK, Tryggvadottir GB. Predictors of quality of life for families of children and adolescents with severe physical illnesses who are receiving hospital-based care. Scand J Caring Sci. 2019 Sep;33(3):698-705. doi: 10.1111/scs.12665. Epub 2019 May 6. PMID 31058346
- [Result] Gotte M, Kesting SV, Winter CC, Rosenbaum D, Boos J. Motor performance in children and adolescents with cancer at the end of acute treatment phase. Eur J Pediatr. 2015 Jun;174(6):791-9. doi: 10.1007/s00431-014-2460-x. Epub 2014 Nov 28. PMID 25428233
- [Result] Sontgerath R, Eckert K. Impairments of Lower Extremity Muscle Strength and Balance in Childhood Cancer Patients and Survivors: A Systematic Review. Pediatr Hematol Oncol. 2015;32(8):585-612. doi: 10.3109/08880018.2015.1079756. Epub 2015 Nov 11. PMID 26558954
- [Result] Baumann FT, Bloch W, Beulertz J. Clinical exercise interventions in pediatric oncology: a systematic review. Pediatr Res. 2013 Oct;74(4):366-74. doi: 10.1038/pr.2013.123. Epub 2013 Jul 15. PMID 23857296
- [Result] Nanthakumar C. The benefits of yoga in children. J Integr Med. 2018 Jan;16(1):14-19. doi: 10.1016/j.joim.2017.12.008. Epub 2017 Dec 14. PMID 29397087
- [Result] Galantino ML, Galbavy R, Quinn L. Therapeutic effects of yoga for children: a systematic review of the literature. Pediatr Phys Ther. 2008 Spring;20(1):66-80. doi: 10.1097/PEP.0b013e31815f1208. PMID 18300936
- [Result] Danhauer SC, Addington EL, Sohl SJ, Chaoul A, Cohen L. Review of yoga therapy during cancer treatment. Support Care Cancer. 2017 Apr;25(4):1357-1372. doi: 10.1007/s00520-016-3556-9. Epub 2017 Jan 7. PMID 28064385
- [Result] Tomlinson D, Diorio C, Beyene J, Sung L. Effect of exercise on cancer-related fatigue: a meta-analysis. Am J Phys Med Rehabil. 2014 Aug;93(8):675-86. doi: 10.1097/PHM.0000000000000083. PMID 24743466
- [Result] Wurz A, Chamorro-Vina C, Guilcher GM, Schulte F, Culos-Reed SN. The feasibility and benefits of a 12-week yoga intervention for pediatric cancer out-patients. Pediatr Blood Cancer. 2014 Oct;61(10):1828-34. doi: 10.1002/pbc.25096. Epub 2014 Jun 17. PMID 24938424
- [Result] Stein E, Rayar M, Krishnadev U, Gupta A, Hyslop S, Plenert E, Schechter-Finkelstein T, Sung L. A feasibility study examining the impact of yoga on psychosocial health and symptoms in pediatric outpatients receiving chemotherapy. Support Care Cancer. 2019 Oct;27(10):3769-3776. doi: 10.1007/s00520-019-04673-9. Epub 2019 Feb 2. PMID 30712097
- [Result] Fukuhara JS, O'Haver J, Proudfoot JA, Spies JM, Kuo DJ. Yoga as a Complementary and Alternative Therapy in Children with Hematologic and Oncologic Disease. J Pediatr Oncol Nurs. 2020 Jul/Aug;37(4):278-283. doi: 10.1177/1043454220909787. Epub 2020 Mar 13. PMID 32167404